CLINICAL TRIAL: NCT06526858
Title: A Prospective, Multicenter, Single Arm, Open-label, Early Feasibility Study to Evaluate Initial Safety and Device Design Concept of "HyperQureTM RDN System", Laparoscopic Renal Denervation Therapy, in Patients With Resistant Hypertension on Three(3) or More Antihypertensive Medications
Brief Title: Early Feasibility Study of "HyperQureTM RDN System", Laparoscopic Renal Denervation Therapy, in Patients With Resistant Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DeepQure Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HQ-HTN-G01
Record Dates: First submitted 2024-07-18; First posted 2024-07-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Resistant Hypertension
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: The HyperQure RDN System consists of a Generator that generates RF(Radiofrequency) energy and a Laparoscopic Instrument that delivers the RF energy generated by the generator to the treatment area. Through a laparoscopic approach, the renal artery is accessed through the retroperitoneum, which is the closest path to the renal artery. After wrapping 360 degrees of renal artery, RDN is performed as per the preset parameters of 50 degrees and 70 seconds. The target blood vessels will be planned by CTA before the procedure, and the proximal and distal areas of the right and left main renal artery are treated once at a distance of at least 3 mm respectively, and RDN will be also performed on the branch or accessory vessels confirmed to be suitable for the RDN procedure by CTA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Extravsacular(Laparoscopic) Renal Denervation (Experimental): Intervention:
  Device: HyperQureTM Renal Denervation (RDN) System:
  * HyperQureTM RDN Generator
  * HyperQureTM RDN Laparoscopic Instrument
  Interventions: Device: HyperQureTM Renal Denervation (RDN) System:

INTERVENTIONS:
Device: HyperQureTM Renal Denervation (RDN) System: — The HyperQure RDN System consists of a Generator that generates RF energy and a Laparoscopic Instrument that delivers the RF energy generated by the generator to the treatment area. Through a extravascular(laparoscopic) approach, the renal artery is accessed through the retroperitoneum, which is the closest path to the renal artery. After wrapping 360 degrees of renal artery, RDN is performed as per the preset parameters of 50 degrees and 70 seconds.
  The target blood vessels will be planned by CTA before the procedure, and the proximal and distal areas of the right and left main renal artery are treated once at a distance of at least 3 mm respectively, and RDN will be also performed on the branch or accessory vessels confirmed to be suitable for the procedure by CTA.
  Other Names: Extravascular renal denervation; Laparoscopic renal denervation

SUMMARY:
HQ-HTN-G01 is a prospective, multicenter, single arm, open label, early feasibility study to evaluate initial safety and device design concept of "HyperQureTM RDN System", laparoscopic renal denervation therapy, in patients with resistant hypertension on three(3) or more antihypertensive medications

DETAILED DESCRIPTION:
<Study purpose> The purpose of this single arm interventional study is to evaluate initial safety and device design concept of HyperQureTM, laparoscopic(extravascular) renal denervation therapy, in patients with resistant hypertension on 3 or more antihypertensive medications including a diuretic The results of this study will be used to 1) prove the concept of complete ablation by Extravascular RDN and 2) develop a solid reference for a pivotal study

<Background and Hypothesis> The HyperQureTM RDN System is developed to overcome the limitations of intravascular RDN using catheters; 1)incomplete renal denervation, 2) risk of endothelial damage due to heat transfer from inside blood vessels by intravascular access, and 3) access limitations due to vascular anatomy and vessel size.

The HyperQureTM RDN System is accessed through the vascular adventitia where renal sympathetic nerves are mainly distributed by retroperitoneal laparoscopic(extravascular) approach . Since the energy is transmitted from outside of vessel by wrapping the blood vessel 360 degrees and the instrument is applicable to small vessels including branch and/or accessory vessels, it is expected that it will be possible to achieve more complete renal denervation, reduce the risk of endothelial damage, and resolve structural access limitations.

<Study plan> Fifteen eligible adult men and women with resistant hypertension will be enrolled and will have Extravascular(laparoscopic) RDN under general anesthesia and will have 36month follow up with various BP evaluations(24hABP, Office BP and Home BP) and CTA/DUS imaging scan evaluations

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to participate if all of the following criteria are met:

1. Aged ≥22 and ≤80 years old at time of enrollment (consent).
2. Diagnosed with resistant hypertension.
3. Office BP ≥140/90 mmHg at Screening Visit 1, and on at least 3 antihypertensive medications of different classes including a diuretic for at least 4 weeks prior to consent.
4. Daytime ABP ≥135/85 mmHg after a four (4)-week run-in period at Screening Visit 2.
5. Agrees to have all study procedures performed, and is competent and willing to provide written, informed consent to participate in this clinical study.

Exclusion Criteria:

Subjects are not eligible to participate if any of the following criteria are met:

1. Has coverage diameter of renal artery less than 2 mm or greater than 11 mm.
2. Has one or more of the following conditions:

   1. Unstable angina with stent implantation (percutaneous coronary intervention) within 3 months of enrolment.
   2. Myocardial infarction within 3 months of enrollment.
   3. Acute heart failure (New York Heart Association (NYHA) III-IV) within 3 months of enrollment
   4. Cerebrovascular accident or transient ischemic attack within 3 months of enrollment.
   5. Atrial fibrillation patients undergoing treatment and not in sinus rhythm. Notes: Patients who have received medical treatment, catheter or surgical treatment for atrial fibrillation and are in sinus rhythm are not excluded
3. Has one or more of the following confirmed anatomical findings in the kidney or renal artery that are not suitable for renal denervation (assessed by the renal CT angiography of Screening 2)

   1. A single functioning kidney.
   2. An atheroma, aneurysm or renal artery stent within 5 mm of the renal denervation site.
   3. Presence of stenosis of 30% or more on all of the blood vessels available for renal denervation therapy.
   4. When it is deemed impossible to perform denervation on both renal arteries according to the discretion of the investigator.
4. Has one or more of the following medical history or a history of surgery/procedure that is not suitable for renal denervation therapy

   1. Renal denervation therapy.
   2. Polycystic kidney disease (PKD).
   3. Atrophic kidney.
   4. Kidney transplant.
   5. Dialysis due to end-stage renal disease.
   6. Any surgery performed on both kidneys. (except endoscopy type of surgery, i.e. endoscopic kidney stone removal)
   7. FMD (Fibromuscular dysplasia)
5. Has comorbidities or surgical/procedural history that are not suitable for retroperitoneal approach

   1. Surgical history through retroperitoneal approach.
   2. Fibrosis in the retroperitoneal region.
   3. Inflammation in the retroperitoneal region.
   4. Severe obesity (body mass index (BMI) > 40 kg/m2)
   5. Risk of increased intracranial pressure
6. Has a history of any intervention for underlying renal artery pathology including stenting or balloon angioplasty.
7. Individual has an eGFR of <45 mL/min/1.73m2, using the 4 variable Modification of Diet in Renal Disease (MDRD) calculation (in mL/min) per 1.73 m2 = 175 x Serum Cr-1.154 x age-0.203 x 1.212 (if patient is black) x 0.742 (if female).
8. Type I diabetes mellitus or uncontrolled Type II diabetes (defined as a plasma Hb1Ac ≥ 9.0%).
9. Has had a reduction of SBP of ≥20 mm Hg or DBP of ≥10 mm Hg within 3 minutes of standing coupled with symptoms during the screening process (at Screening Visit 2).
10. Requires chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea (e.g., CPAP, BiPAP).
11. Has documented primary pulmonary hypertension.
12. Has an untreated secondary cause of hypertension (either known or suspected) or is taking drugs that increase sympathetic tone and could contribute to hypertension.
13. Has a scheduled or planned surgery that, in the opinion of the Investigator, may affect study endpoints.
14. Works night shifts.
15. Has severe cardiac valve stenosis for which, in the opinion of the Investigator, a significant reduction of blood pressure is contraindicated.
16. Is pregnant, nursing or planning to become pregnant during the course of the study follow-up (Note: Female participants of childbearing potential must have a negative serum or urine human chorionic gonadotropin (hCG) pregnancy test prior to angiography).
17. Has a known unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable, in the opinion of the Investigator, to comply with study follow-up requirements.
18. Has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
19. Patients who are at high risk if taken off their anticoagulant and antiplatelet agents for a few days.
20. Allergy, intolerance or contraindications to contrast medium.
21. Prescribed any standard antihypertensive cardiovascular medication for other chronic conditions (e.g. ischemic heart disease) for less than 90 days before Screening visit 1 and whose discontinuation might pose serious risk to health.
22. Has frequent intermittent or chronic pain that results in the treatment with non-steroidal anti-inflammatory drugs (NSAIDs) for two (2) or more days per week over the month prior to Screening Visit 2.
23. Concurrent enrollment in any other investigational drug or device study(Participation in non-interventional Registries is acceptable).

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2029-03-20 (Estimated)

PRIMARY OUTCOMES:
Decrease in 24-h Ambulatory Systolic Blood Pressure(ASBP) | from baseline to 3 months post procedure
  Measure by 24-hour ambulatory blood pressure monitoring(ABPM)
• Incidence of major adverse events (MAE). Defined as a composite of the following events, through 1-month post-procedure | from baseline to1-month post-procedure
  * All-cause mortality.
  * End-stage renal disease (ESRD).
  * Significant embolic event resulting in end-organ damage
  * Renal artery perforation requiring intervention.
  * Renal artery dissection requiring intervention.
  * Vascular complications.
  * Injury to surrounding structures (inc. vasculature structure, the ureters, colon and or other intraabdominal and/or retroperitoneal structures).
  * Hospitalization for hypertensive crisis not related to confirmed nonadherence with medications or the protocol.
  * New renal artery stenosis >70%, as diagnosed by DUS and confirmed by Computed Tomography Angiogram (CTA) or diagnosed/confirmed by renal CTA.
  * Prolongation of hospitalization after the index intervention for device or procedural related issues.
  * Major bleeding (bleeding Type 3a or higher according to the Bleeding Academic Research Consortium [BARC]2; overt bleeding plus a hemoglobin drop of 3 to 5 g/dL; any transfusion with overt bleeding).

SECONDARY OUTCOMES:
Change in 24-h ASBP | from baseline to 6-, 12-, 24-, 36-months post procedure.
  Measure by 24-hour ambulatory blood pressure monitoring(ABPM)
Change in 24-h Ambulatory Diastolic Blood Pressure(ADBP) | from baseline to 3-, 6-, 12-, 24-, 36-months post procedure.
  Measured by 24-hour ABPM
Change in daytime ASBP and ADBP | from baseline to 3-, 6-, 12-, 24-, 36-months post procedure
  Measured by 24 hour ABPM
Change in nighttime ASBP and ADBP | from baseline to 3-, 6-, 12-, 24-, 36-months post procedure
  Measured by 24 hour ABPM
Change in Office Systolic Blood Pressure(SBP) and Diastolic Blood Pressure(DBP) | from baseline to 1-, 3-, 6-, 12-, 24-, 36-months post-procedure
  Measured by Office BP device
Change in Home Systolic Blood Pressure(SBP) and Diastolic Blood Pressure(DBP) | from baseline to 1-, 3-, 6-, 12-months post procedure
  Measured by Home BP device
Incidence of achieving target office SBP (SBP <140 mmHg) | from baseline to 1-, 3-, 6-, 12-, 24-, 36-months post-procedure
  Number of achieving target office SBP measured by Office BP device
Incidence of each of the following acute/procedural adverse event | from baseline to 1-month post-procedure
  * Procedural complication (≥grade 3) as per Clavien-Dindo classification.
  * Significant embolic event resulting in end-organ damage.
  * Renal artery perforation requiring intervention.
  * Renal artery dissection requiring intervention.
  * Vascular complications.
  * ESRD.
  * ≥40% decline in estimated glomerular filtration rate (eGFR).
  * New myocardial infarction.
  * New stroke.
  * Renal artery re-intervention.
  * Increase in serum creatine >50% from Screening Visit 2.
  * Hospitalization for hypertensive crisis not related to confirmed nonadherence with medications or the protocol.
  * New renal artery stenosis >70%, diagnosed by DUS and confirmed by computed tomography (CT) angiography or diagnosed/confirmed by CTA.
Incidence of each of the following chronic adverse event | from baseline to 3-, 6-, 12-, 24-, 36-months post-procedure
  * All-cause mortality.
  * ESRD (≥40% decline in eGFR).
  * New myocardial infarction.
  * New stroke.
  * Renal artery re-intervention.
  * Increase in serum creatine >50% from Screening Visit 2.
  * Hospitalization for hypertensive crisis not related to confirmed nonadherence with medications or the protocol.
  * New renal artery stenosis >70%, diagnosed by DUS and confirmed by CT angiography or diagnosed/confirmed by CTA

OTHER OUTCOMES:
Change in antihypertensive medication usage | from baseline up to 36-months post procedure
  Medication change(number, type, dose) will be evaluated by drug surveillance diary and blood/urine drug testing

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California Irvine, Orange, California
  - Stanford Health Care, Stanford, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Henry Forth Health, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No